CLINICAL TRIAL: NCT04020315
Title: Effect of Non-surgical Periodontal Treatment on GCF HIF-1α, VEGF and TNF-α Levels in Generalized Aggressive Periodontitis Patients.
Brief Title: GCF HIF-1α, VEGF and TNF-α Levels in G-AgP Patients Before and After Periodontal Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Beral Afacan, Principal Investigator, Aydin Adnan Menderes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AggressiveHIF
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Aggressive Periodontitis, Generalized; Periodontal Health
Keywords: aggressive periodontitis; gingival crevicular fluid; hypoxia; cytokines
MeSH Terms: conditions — Aggressive Periodontitis; Hypoxia | interventions — Root Planing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Generalized aggressive periodontitis (Experimental): Non-surgically performed scaling and root planing.
  Interventions: Procedure: Non-surgically performed scaling and root planing

INTERVENTIONS:
Procedure: Non-surgically performed scaling and root planing — Non-surgically performed scaling and root planing

SUMMARY:
Hypoxia-inducible angiogenic pathway involving hypoxia inducible factor-1 alpha (HIF-1α), vascular endothelial growth factor (VEGF) and tumour necrosis factor- alpha (TNF-α) may regulate the several biological processes related to inflammation. Generalized aggressive periodontitis (G-AgP) is a rare but highly destructive form of inflammatory periodontal disease. The present study aimed to assess the effect of non-surgical periodontal treatment on gingival crevicular fluid (GCF) HIF-1α, VEGF and TNF-α levels in G-AgP patients. 20 G-AgP and 20 periodontally healthy subjects were enrolled. At baseline, GCF samples were collected and whole mouth clinical periodontal parameters were recorded. G-AgP patients received non-surgical periodontal treatment. Clinical parameters and GCF cytokines were re-measured at 1 and 3 months after treatment. GCF HIF-1α, VEGF and TNF-α levels were analyzed by ELISA. Data were analyzed using appropriate statistical tests.

DETAILED DESCRIPTION:
Study Population and Clinical Examination

A total of 40 individuals were recruited for the present study. Inclusion criteria included: 1) aged 25 to 45 years 2) non-smokers with no history of smoking 3) having at least 20 natural teeth. Exclusion criteria were as follows: 1) having any diagnosed medical disorders such as diabetes mellitus, cardiovascular diseases, rheumatoid arthritis, immunological and mucocutaneous diseases 2) usage of antibiotics, non-steroidal anti-inflammatory drugs and immunosuppressive agents within the past 6 months 3) having any non-inflammatory destructive periodontal disease 4) nonsurgical/surgical periodontal therapy received in the past year 5) having a restorative and endodontic treatment requirement 6) having orthodontic appliances or a removable partial denture 7) pregnant/ lactating/ postmenopausal females.

The whole mouth clinical periodontal examination included measurement of probing depth (PPD), clinical attachment level (CAL), presence of bleeding on probing (BOP), gingival index (GI) and plaque index (PI) at 6 sites per tooth, except the third molars. The presence and type of the alveolar bone loss were assessed on the digital panoramic radiograph in each participant, which was supplemented with periapical radiographs if necessary.

Periodontal status of each patient was evaluated by a single calibrated periodontists with a manual probe. The diagnosis of G-AgP or periodontally health was determined according to the International Classification of Periodontal Diseases in 1999. The patients in G-AgP group (n=20) had a minimum three teeth apart from the first molars and incisors showing CAL ≥5 mm and PPD ≥6 mm. Radiographic bone loss was ≥30 % of root length affecting ≥3 teeth other than first molars and incisors. This generalized pattern of severe destruction was inconsistent with the amount of microbial deposits. Patients had at least one other family member presenting with or having a history of severe periodontal problems. Periodontally healthy individuals (n=20) in the control group had no sites with PPD >3 mm and CAL >2 mm and also no radiographic evidence of alveolar bone loss. BOP was <15% in the whole mouth.

Treatment

The recruited G-AgP patients received conventional quadrant scaling and root planning (SRP) under local anaesthesia for 3 weeks. SRP was performed by the same periodontist (who was different the investigator recorded periodontal parameters) using ultrasonic inserts and manual periodontal curettes. Re-evaluations were performed at 1 and 3 months following the completion of the SRP in the lower right quadrant. No periodontal intervention was carried out in the periodontally healthy controls.

GCF sampling

GCF was sampled from two deepest pockets of single-rooted teeth at baseline in G-AgP group immediately before the treatment of upper right quadrant. Sampling was repeated at the same sites following the completion of the SRP in the lower right quadrant. GCF was sampled from the buccal aspects of two nonadjacent interproximal sites in single-rooted teeth with. Samples were collected from the sites without BOP in the periodontally healthy group. Standardized filter paper strips were used for GCF sampling. Sterile paper strips were gently inserted into the gingival sulcus or pocket until mild resistance was felt and left there for 30 s. The absorbed fluid volume was measured with a precalibrated electronic device. The paper strips were stored at -40◦C for further analysis.

Measurement of HIF-1α, VEGF and TNF-α Levels in GCF

Two paper strips were pooled, placed in 300 µL PBS-T (0.05%). HIF-1α, VEGF and TNF-α levels in GCF samples were measured by the enzyme-linked immunosorbent assay using commercial kits in line with the manufacturer's guidelines. GCF results were expressed as both total amounts at two sites per sampling time.

Statistical Analysis

All statistical analyses were carried out with the standard statistical software package. For the intra-group comparisons, if the data were not normally disturbed, Friedman test and the Dunn test with the Bonferroni correction were used to analyze the change between baseline and 1 month and 3 months after treatment. For inter-group comparisons, Mann-Whitney U test for normally and non-normally disturbed data. The Spearman's rank correlation test was used to detect the correlations of biochemical parameters with clinical parameters and each others in diseased group before and after treatment. All tests were performed at significance level of P <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. aged 25 to 45 years
2. non-smokers with no history of smoking
3. having at least 20 natural teeth.

Exclusion Criteria:

1. having any diagnosed medical disorders such as diabetes mellitus, cardiovascular diseases, rheumatoid arthritis, immunological and mucocutaneous diseases
2. usage of antibiotics, non-steroidal anti-inflammatory drugs and immunosuppressive agents within the past 6 months
3. having any non-inflammatory destructive periodontal disease
4. nonsurgical/surgical periodontal therapy received in the past year
5. having a restorative and endodontic treatment requirement
6. having orthodontic appliances or a removable partial denture
7. pregnant/ lactating/ postmenopausal females.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Gingival crevicular fluid protein content change | Change from baseline to 1 month and 3 months after treatment
  pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University, Faculty of Dentistry, Department of Periodontology, Aydin, Turkey (Türkiye)